CLINICAL TRIAL: NCT07199413
Title: Allogeneic, Antigen-Presenting, GM-CSF-secreting, SV-BR-1-GM Whole Cell-Therapeutic Vaccine and Immunotherapy: A Phase I Pilot Safety and Feasibility Study for Solid Tumor Patients With CNS Metastases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sailaja Kamaraju, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-KAMARAJU-ASTRO
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; Leptomeningeal Metastasis
Keywords: solid tumor patients; CNS Metastases; SV-BR-1-GM Vaccine; Immunotherapy
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — Cyclophosphamide; pembrolizumab; Interferons; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccine and Study Drugs (Experimental)
  Interventions: Biological: SV-BR-1-GM Vaccine; Drug: Cyclophosphamide; Drug: Pembrolizumab; Drug: Interferon

INTERVENTIONS:
Biological: SV-BR-1-GM Vaccine — ~20 X 10^6 cells across 4 injection sites
Drug: Cyclophosphamide — 300 mg/m^2 Intravenous
  Other Names: Cytoxan
Drug: Pembrolizumab — 200 mg/m^2 Intravenous
  Other Names: Keytruda
Drug: Interferon — 0.18 mcg subcutaneous
  Other Names: Sylatron

SUMMARY:
This is a prospective, single-center, phase 1 basket trial that will evaluate the safety and feasibility of administering SV-BR-1-GM in combination with pembrolizumab to solid tumor oncology patients over nine cycles.

DETAILED DESCRIPTION:
This prospective, single-site, open-label, single-arm, phase 1 basket trial is designed to evaluate whether a SV-BR-1-GM vaccine and pembrolizumab combination therapy is safe and can be feasibly administered to solid cancer patients with brain metastases who progress on SOC therapy. Secondary objectives will determine the preliminary efficacy of the study regimen, while exploratory measurements will evaluate underlying mechanisms and biomarkers of response using patient biospecimens (peripheral blood and, when available, CSF). A total of 20 solid tumor oncology patients, accrued over a 24-month time period, will be treated with the SV-BR-1-GM vaccine and pembrolizumab over nine three-week cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subject has a prior diagnosis of central nervous system (CNS) metastases per institutional standard of care and/or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria on imaging.
3. Subject has disease progression of CNS metastases (brain and/or leptomeningeal metastases (LMD) ) with progression on ≥ 1 line of standard of care therapy.
4. Patients should have at least one metastasis approved by the research team that meets the following size requirements:

   o Diagnosis and treatment response to measurable CNS and LMD will be per institutional and/or RANO-BM criteria modified to include the cut off point of 0.5 cm or higher.
   1. Patients with recurrent and or progressive symptomatic or asymptomatic brain lesions and >0.5 cm and twice the magnetic resonance imaging (MRI) slice thickness are allowed.
   2. Any recurrent or progressive brain lesions > 3 cm in size and or causing symptoms must be evaluated by the study team for SRC and or whole brain radiation therapy (WBRT) prior to study entry.
   3. Patients with recurrent brain lesions that are not treatable with local therapy or WBRT are eligible.
   4. An interval of at least 4 weeks after the end of whole brain radiation or for any surgical resection of brain lesions is permitted; an interval of at least 4 weeks or 5 half-lives (whichever is sorter) after the last cytotoxic, targeted, immunotherapeutic or investigational agent is permitted (prior to the start of DC vaccine).
   5. Patients should have recovered from the AEs of prior therapy to baseline or Grade ≤ 1.
   6. Patients with recurrent or progressive LMD are eligible.
5. Prior surgical resection of the brain metastases is allowed; patients must recover for at least four weeks prior to study enrollment.
6. Patients with extracranial disease are eligible as long as no signs of visceral crisis.
7. Prior immunotherapy is allowed.
8. No need for steroids for at least two weeks.

   1. Patients who recently started steroids should have completed tapering to be eligible.
   2. Patients who have been on chronic steroids are eligible as long as they are maintained on a dose of ≤ 10 mg of prednisone or equivalent.
9. Tumor not impinging on the middle cerebral artery/speech-motor strip.
10. Patients who undergo any other surgical procedures (other than SRS) must have recovered for at least 3-4 weeks before study entry.
11. Subject has a life expectancy of ≥ 12 weeks.
12. ECOG 0-2.
13. Preserved organ function.

    1. ANC ≥ 1,000/µl
    2. Platelets ≥ 10,000 µl
    3. Hemoglobin ≥ 8 gm/dL
    4. Bilirubin ≤ 1.5 mg/dL; those with Gilbert syndrome may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN.
    5. Creatinine clearance ≥ 50 mL/min
    6. AST, ALT ≤ 2.5 times institutional upper limit
    7. ALP ≤ 2.5 × institutional upper limit, with the exception that ALP of < 5 x ULN is acceptable in patients with elevated ALP due to bone metastases (in the absence of liver metastases).
14. Patients with lymphopenia are eligible at the discretion of the treating provider.
15. Female subjects must meet one of the following:

    1. Postmenopausal for at least one year before enrollment, or surgically sterile (i.e., undergone bilateral oophorectomy).
    2. Premenopausal is defined as someone who has had menses at any time in the preceding 12 months. Premenopausal women who are eligible for this trial will require a GnRH analogue and treating physician, per institutional guidelines, may choose to monitor the ovarian function with laboratory tests (FSH/LH/Estradiol) to ensure a complete menopausal status with cessation of menses.

    i. Note: Pregnancy test should be administered per institutional guidelines.
16. Male patients must be willing to abstain from heterosexual activity and/or use a condom during treatment and three months after treatment discontinuation.
17. Willing to provide blood for biomarker assessments.
18. Optional CSF, when appropriate, for biomarker assessments (at the discretion of treating physician).
19. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. History of allergic reactions or intolerance to immunotherapy.
2. History of active or untreated infection, such as chronic untreated infections, HIV, Hepatitis B, Hepatitis C, or tuberculosis.
3. History of active inflammatory or autoimmune disease (granulomatosis, polyangiitis, Graves' disease, rheumatoid arthritis, polyphisitis, uveitis, etc.), except for the following.

   1. Vitiligo; alopecia
   2. Hypothyroidism: stable on replacement therapy
   3. Chronic skin disease that doesn't require steroid therapy.
   4. Active celiac disease or inflammatory bowel disease
4. Presence of severe neurological symptoms and unable to participate in the study due to acute decompensation.
5. History of severe brain injury.
6. History of last dose of antineoplastic therapy ≤ 7 days prior to the first dose of study drug. If sufficient wash-out time has not occurred (defined as 5 half-lives of the prior antineoplastic therapy), a longer wash-out may be needed, as suggested by the study team.
7. Patients with myelodysplastic syndrome (MDS), leukemia, or active blood disorders.
8. Patients with prior history of poorly controlled diabetes, lung disease, primary immunodeficiency syndromes.
9. Severe cardiac disease as determined by the treating providers.
10. Life expectancy <12 weeks.
11. Acute spinal cord compression, unless considered to have received definitive treatment for this and clinical evidence of stable disease for at least 28 days.
12. Active treatment with prednisone >10 mg or equivalent steroid (e.g., >1.5 mg dexamethasone) per day and/or other immunosuppressive therapies (e.g., interferon, azathioprine, mycophenolate).
13. Presence of secondary malignancies (chronic lymphocytic leukemia [CLL], and other hematological or solid tumor malignancies), with the exception of in situ disease (ductal carcinoma in situ [DCIS], lobular carcinoma in situ [LCIS], cervical intraepithelial neoplasia [CIN], squamous cell and basal cell cancer, or remote history of successfully treated melanoma).
14. Active participation in other clinical trials evaluating an active investigational drug within the past four weeks.
15. Unresolved toxicities of NCI CTCAE Grade ≥ 2 such as neurotoxicity, cardiotoxicity, myelotoxicity, gastrointestinal, or others.
16. Patients who received prior immune checkpoint inhibitors (CPIs) and have not recovered from Grade ≥ 2 AEs related to CPIs.
17. Women of childbearing potential who do not agree to precautions outlined in the inclusion criteria or having positive pregnancy tests.
18. Men who are sexually active and not willing to use effective contraceptives (e.g., condoms) during and 3 months after treatment.
19. Women who are pregnant or nursing.
20. Severe mental illness per physician's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or higher adverse events | 30 days after the beginning of study therapy, 9 months after the beginning of study therapy
  The number of grade 3 or higher adverse events (AEs). AEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse (CTCAE), version 5.0.
Study therapy duration | 6 months
  The number of subjects who complete six months of the investigational agent (vaccine).

IPD SHARING:
Plan to Share IPD: No